CLINICAL TRIAL: NCT01887834
Title: The Effect of Kyo-Dophilus 1.5 Billion on the Symptoms of Severe Irritable Bowel Syndrome
Brief Title: Efficacy of a Multi-strain Probiotic in the Treatment of Irritable Bowel Syndrome
Acronym: IBS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry); Dicentra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1302
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome; Digestive System Diseases; Colonic Diseases, Functional; Colitis, Mucous; Colon, Irritable
Keywords: bloating; constipation; diarrhea; gas; mucous; cramping
MeSH Terms: conditions — Irritable Bowel Syndrome; Digestive System Diseases; Colonic Diseases, Functional; Constipation; Diarrhea; Mucopolysaccharidosis IV; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kyodophilus matching placebo capsules (Placebo Comparator): Kyodophilus Matching Placebo Capsules
  Subjects will be provided with two bottles containing 30 capsules each of matching placebo upon randomization. Subjects will be instructed to take one capsule with breakfast daily for the full 12 weeks duration of the trial. While one bottle contains enough capsules for the time frame between each visit, two bottles have been provided to permit a surplus in the event scheduling conflicts arise. The third bottle, providing the remainder or study capsules, will be provided at visit 2.
  Interventions: Dietary Supplement: Kyodophilus Matching Placebo Capsules
- Kyodophilus multi strain probiotic capsules (Active Comparator): Kyodophilus multi-strain probiotic capsules
  The Kyo-Dophilus study product is a gelatin capsule containing three proprietary probiotic bacterial strains. The total quantity of bacteria per capsule is 1.5 billion colony forming units (1.5 x 109 cfu) and is composed of the following strains:
  * Lactobacillus gasseri KS-13 1.2
  * Bifidobacterium bifidum G9-1 0.15
  * Bifidobacterium longum MM-2 0.15
  Subjects will be provided with two bottles containing 30 capsules each of matching placebo upon randomization. Subjects will be instructed to take one capsule with breakfast daily for the full 12 weeks duration of the trial. While one bottle contains enough capsules for the time frame between each visit, two bottles have been provided to permit a surplus in the event scheduling conflicts arise. The third bottle, providing the remainder or study capsules, will be provided at visit 2.
  Interventions: Dietary Supplement: Kyodophilus multi-strain probiotic capsules

INTERVENTIONS:
Dietary Supplement: Kyodophilus multi-strain probiotic capsules
  Arms: Kyodophilus multi strain probiotic capsules
Dietary Supplement: Kyodophilus Matching Placebo Capsules
  Arms: Kyodophilus matching placebo capsules

SUMMARY:
The Canadian College of Naturopathic Medicine is conducting a research study on Irritable Bowel Syndrome (IBS), a common condition in North America. It is a long term, recurring gastrointestinal disorder that is estimated to affect 30% of the general population. IBS is characterized by abdominal pain and cramps, and bowel dysfunction such as diarrhea and bloating.

The medicines that are currently used to help people with IBS are not as effective as we would like them to be. These medicines are usually only prescribed to reduce the pain of IBS and not actually treat the disorder itself. Recently, scientists have found that probiotics (beneficial bacteria that live inside humans) may help reduce the painful symptoms and diarrhea that are part of IBS.

This research is being conducted to determine whether this particular combination of three probiotic bacteria (named Lactobacillus gasseri, Bifidobacterium bifidum and Bifidobacterium longum) will reduce the symptoms of severe IBS.

DETAILED DESCRIPTION:
The purpose of this trial is to investigate the effects of the three strain probiotic, Kyo-Dophilus, on the symptoms associated with severe Irritable Bowel Syndrome. A previous pilot clinical trial identified individuals with severe IBS to be most likely to benefit from the treatment provided in this trial.

The primary objective of this trial is to determine the effectiveness of Kyo-Dophilus on the symptoms associated with Irritable Bowel Syndrome in an adult population diagnosed with Irritable Bowel Syndrome by ROME III criteria and classified as severe through the Irritable Bowel Severity Scoring System and to measure quality of life and global well-being of patients through the Adequate Relief Criteria and the Irritable Bowel Syndrome-Quality of Life Questionnaire.

The secondary objective is to assess the tolerability of the treatment through the use of Adverse Event Reporting Forms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18-64.
* A diagnosis of Irritable Bowel Syndrome as per ROME III criteria.
* A classification of severe irritable bowel syndrome as indicated by the Irritable Bowel Severity Scoring System (score >300).
* Female subjects currently using an acceptable form of birth control who agree to maintain its use throughout the study (e.g. abstinence, oral contraceptives, barrier methods).
* Subjects who agree to maintain their current eating habits throughout the study.
* Ability to understand and sign the Informed Consent Form.

Exclusion Criteria:

* Female subjects who are breastfeeding, pregnant, or are open to becoming pregnant in the next three months
* Subjects currently receiving medication for the treatment of IBS symptoms.
* Subjects currently receiving natural health products for treatment of IBS symptoms will be eligible for inclusion in the trial is they agree to undergo a four week washout period.
* Subjects currently experiencing nausea, fever, vomiting, bloody diarrhea or severe abdominal pain.
* Subjects who are immune-compromised (e.g. AIDS, lymphoma, patients undergoing long-term corticosteroid treatment).
* Subjects currently receiving antibiotic therapy or antibiotic therapy within the previous month.
* Subjects regularly (>3 times weekly) consuming probiotics enriched products (e.g. probiotic enriched yogurts, Activia, etc…).
* Subjects who have recently (< 3 months) initiated dietary measures to control IBS symptoms, such as elimination of certain foods.
* Subjects with a history of major or complicated gastrointestinal surgery.
* Subjects with severe endometriosis.
* Subjects with malignant tumors or subjects undergoing chemotherapy or radiation therapy.
* Subjects with severe IBS that require medication for treatment of IBS symptoms.
* Subjects with weight loss, anemia, inflammatory bowel disease, or celiac sprue, and family history of colorectal cancer.
* Subjects exhibiting or indicating thoughts of suicide currently or in the past as based on patient screening interview by the investigator/clinician. Appropriate referral to a health care provider will be provided.
* Subjects with known allergies to milk or milk based products.
* Subjects using and/or have used antipsychotic or anticholinergic medication within the prior month, those with reported significant abnormalities on thyroid function tests, blood counts and serum chemistry.
* Subjects 50 years or older who have been diagnosed with IBS and have not received a colonoscopy in the last five years.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Severity | 12 weeks
  Irritable bowel severity scoring system is a validated questionnaire used to monitor IBS (Francis et al, 1997).

SECONDARY OUTCOMES:
Tolerability of the treatment | 12 weeks
  A standardized Adverse Events Reporting Form will be used to query subjects on the incidence of any side effects, which will be recorded.

OTHER OUTCOMES:
The Irritable Bowel Syndrome-Quality of Life Questionnaire | 12 weeks
  This is a validated quality of life questionnaire (Patrick et al, 1998)
Adequate Response Criteria | 12 weeks
  The Adequate Response criteria assesses the overall clinical relevance of the intervention under investigation: e.g. "In the past 7 days, have you had adequate relief (AR) of your IBS pain and discomfort?" (Ko et al, 2011; Guglielmetti et al, 2011; Ligaarden et al, 2010; Sondergaard et al, 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Dugald Seely, ND, Principal Investigator — The Canadian College of Naturopathic Medicine
Locations (1):
- The Canadian College of Naturopathic Medicine, Toronto, Ontario, Canada